CLINICAL TRIAL: NCT03610867
Title: A Phase I, Randomized, Double-blind, Placebo Controlled, Ascending Dose Study in Healthy Chinese Volunteers to Evaluate the Safety, Tolerability, and Pharmacokinetics (PK) Profile of Single and Multiple Ascending Oral Doses of TG-2349
Brief Title: To Evaluate the Safety, Tolerability, and Pharmacokinetics Profile in Healthy Chinese Volunteers of TG-2349
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dongguan HEC TaiGen Biopharmaceuticals Co., Ltd. (Industry)
Collaborators: R&G Pharma Studies Co.,Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: TG-2349-C-01
Record Dates: First submitted 2018-05-06; First posted 2018-08-01 (Actual); Last update posted 2018-08-02 (Actual); Status verified 2018-08

CONDITIONS: Healthy Chinese Volunteers
Keywords: safety; tolerability; PK; single ascending oral dose; multiple ascending oral doses
MeSH Terms: interventions — Sagittal Abdominal Diameter; mycophenolic adenine dinucleotide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Furaprevir capsule (SAD) (Experimental): single ascending oral dose (100 mg, 200 mg, 400 mg, and 600 mg) of TG-2349 (Furaprevir capsule)
  Interventions: Drug: Furaprevir capsule (SAD)
- Placebo (SAD) (Placebo Comparator): Single ascending oral dose of Furaprevir similar capsule.
  .
  Interventions: Drug: Placebo (SAD)
- Furaprevir capsule (MAD) (Experimental): multiple ascending oral doses (200 mg, 400 mg, and 600 mg) of TG-2349 (Furaprevir capsule)
  Interventions: Drug: Furaprevir capsule (MAD)
- Placebo (MAD) (Placebo Comparator): Multiple ascending oral doses of Furaprevir similar capsule
  Interventions: Drug: Placebo (MAD)

INTERVENTIONS:
Drug: Furaprevir capsule (SAD) — There are four doses in this part, 100 mg, 200 mg, 400 mg, and 600 mg. Each subject will receive the sample once by oral administration.
  Other Names: TG-2349 (SAD)
  Arms: Furaprevir capsule (SAD)
Drug: Furaprevir capsule (MAD) — There are three doses in this part, 200 mg, 400 mg, and 600 mg. Each subject will be allocated into one dosing regimen and receive the sample once daily for 5 consecutive days by oral administration.
  Other Names: TG-2349 (MAD)
  Arms: Furaprevir capsule (MAD)
Drug: Placebo (SAD) — Each subject will receive the sample once by oral administration.
  Arms: Placebo (SAD)
Drug: Placebo (MAD) — Each subject will be allocated into one dosing regimen and receive the sample once daily for 5 consecutive days by oral administration.
  Arms: Placebo (MAD)

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and pharmacokinetics (PK) profile of different doses of TG-2349 (Furaprevir capsule) in healthy Chinese volunteers.

DETAILED DESCRIPTION:
This study is to evaluate the safety, tolerability, and pharmacokinetics (PK) profile in healthy Chinese volunteers with single or multiple ascending oral doses of TG-2349 (Furaprevir capsule). The study is separated into two parts, part A and part B.

Part A：To evaluate the safety, tolerability, and PK profile of single ascending oral dose (100 mg, 200 mg, 400 mg, and 600 mg) of TG-2349 in healthy Chinese volunteers.

Part B：To evaluate the safety, tolerability, and PK profile of multiple ascending oral doses (200 mg, 400 mg, and 600 mg) of TG-2349 for five days in healthy Chinese volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Before starting the study, an informed consent form (ICF) approved by the Institutional Review Board (IRB) is obtained from the subject or his/her legal representative；
2. Male or female, and 18 to 45 years of age inclusive when signing ICF；
3. Body mass index (BMI) in the range of 19.0 to 24.0 kg/m2 and male body weight ≥ 50 kg, female body weight ≥ 45 kg；
4. In generally good physical and mental health status on basis of a medical history review, physical examination and vital signs, 12-lead ECG, and laboratory results at screening；
5. For females, one of the following criteria must be fulfilled

   1. Had undergone surgical sterilization, or
   2. Subjects of childbearing potential must satisfy the following criteria:

   Before group assignment, the pregnancy test is negative, and Subjects agree to use an approved contraceptive method (i.e. oral spermicidal agent, condoms, or intrauterine devices) during the entire study period (from signing ICF to the last visit). Subjects must also consent to keep the contraceptive method unchanged until 1 month after the study, and Breastfeeding is prohibited
6. Males must be willing to use a reliable form of contraception (use of a condom or spouses using any of the above standards) during the entire study period (from signing ICF to the last visit)；
7. Have not used tobacco or nicotine-containing products within 1 month prior to the first dose of study drug；
8. Have not drunk alcohol beverages or drank alcoholic beverages less than 12 times within 3 months prior to the first dose of study drug；
9. Willing to abstain from caffeine- or xanthine-containing beverages, including coffee and tea, chocolate, alcohol, grapefruit juice, and Seville oranges juice before 24 hr and during the Stay-on Site period.

Exclusion Criteria:

1. Current, prior history, or family history of any disease of sudden cardiac death, myocardial ischemia, myocardial infarction, congestive heart failure, QT prolongation syndrome, hypokalemia, myocarditis, exertional dyspnea, cerebrovascular injury, venous thromboembolism；
2. Requires concomitant medication associated with increased QTc interval (i.e. Class I or III antiarrhythmic agents or with cardiac insufficiency；
3. Any abnormality on 12-lead ECG: PR>240 ms, PR<110 ms, QRS>110 ms, QTc>450 ms, or bradycardia ( heart rate < 50 beats/min) at screening or the day -1；
4. Any clinical significant abnormality on 12-lead ECG (i.e. atrioventricular block, TdT, other types of ventricular tachycardia, atrial fibrillation and ventricular flutter, clinical significant abnormality on T wave changes or any abnormality on 12-lead ECG that effects QTc intervals) at screening or the day -1；
5. Systolic pressure>140 mmHg or <90 mmHg, diastolic pressure >90 mmHg, pulse <50 beats/min or >100 beats/min at screening or the day -1；
6. Any clinical significant abnormality on chest X-rays or abdominal ultrasound scan at screening；
7. Positive serological test for hepatitis A (IgM anti-HAV), hepatitis B (HbsAg), hepatitis C (anti-HCV antibody), or syphilis at screening；
8. Pregnant or breastfeeding；
9. Any abnormal laboratory values (normal value ±10％) that are considered clinical significant by the Investigator at screening or the day -1；
10. Positive breath alcohol test or urine drug screen at screening or the day -1；
11. Current or prior history of any disease of diabetes, cardiovascular, hepatic or renal impairment；
12. Any malabsorption syndrome or other gastrointestinal disturbances affecting drug absorption；
13. Difficulty with blood collection and/or poor venous access for the purposes of phlebotomy；
14. History of epileptic seizure, mental disorders affecting the subject's compliance with the protocol, suicidal risk, or a history of alcohol or illicit drug abuse；
15. Currently has any disease that seriously affects the immune system, for instance, human immunodeficiency virus (HIV) infection, hematological malignancy, solid cancer or splenectomy；
16. Allergy, hypersensitivity or allergic reaction to Furaprevir or its excipients, or Sulfonamides；
17. History of surgery within 6 months prior to the first dose of study drug；
18. Received any hepatic enzyme inducers or hepatic enzyme inhibitors within 30 days prior to the first dose of study drug through medical history questionnaire (refer to appendix 2)；
19. Received any investigational drugs within 3 months prior to the first dose of study drug；
20. Received any prescription drugs, over-the-counter (OTC) drug, or Chinese herbal medicines within 14 days prior to the first dose of study drug；
21. Received any nutritional supplies, including multivalent cations products (i.e. Ca-, Al-, Mg-, Fe-, and Zn-containing products, sucralfate, antacid, nutritional supplements, multi-vitamin, supplements for metals) within 7 days prior to the first dose of study drug；
22. Blood donation ≥400 ml within 3 months prior to the first dose of study drug；
23. Any disease or situation that would affect the safety of study drug or pharmacokinetics profile by Investigators' judgments；
24. As determined by Investigator, a subject is not suitable to take part in this study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2017-04-27 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
Cmax (Maximum Plasma Concentration) | 10 days
  Maximum Plasma Concentration
Tmax (Time at Which Maximum Plasma Concentration is Observed) | 10 days
  Time at Which Maximum Plasma Concentration is Observed
AUC (Area Under the Plasma Concentration) | 10 days
  Area Under the Plasma Concentration
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 10 days
  CTCAE v4.0

SECONDARY OUTCOMES:
12-lead ECG (electrocardiogram) | 10 days
blood pressure (mmHg) | 10 days
  Vital signs
pulse (beats/ min) | 10 days
  Vital signs
respiratory rate (breaths/ min) | 10 days
  Vital signs
body temperature (oC) | 10 days
  Vital signs
General Appearance Physical examination | 10 days
  Physical examination
Skin Physical examination | 10 days
  Physical examination
Head and Neck Physical examination | 10 days
  Physical examination
Chest region Physical examination | 10 days
  Physical examination
Abdominal region Physical examination | 10 days
  Physical examination
Back region Physical examination | 10 days
  Physical examination
Extremities Physical examination | 10 days
  Physical examination

CONTACTS AND LOCATIONS:
Overall Officials: Pingsheng Xu, PhD, Principal Investigator — Xiangya Hospital of Central South University
Locations (1):
- Xiangya Hospital Central South University, Changsha, Hunan, China